CLINICAL TRIAL: NCT06800768
Title: The Value of 68Ga-FAPI PET/CT in Detecting Recurrent and Metastatic Lesions in Patients with Thyroid Cancer After Surgery
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hu Jiajia, Deputy director, Ruijin Hospital
Other Study IDs: RuijinH 2025-15
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Thyroid Cancer
Keywords: Thyroid Cancer; 68Ga-FAPI; PET/CT
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with suspected recurrence or metastasis of thyroid cancer after surgery

SUMMARY:
This study aims to investigate the value of 68Ga-FAPI PET/CT in detecting recurrent and metastatic lesions in patients with thyroid cancer after surgery.

DETAILED DESCRIPTION:
The investigators will number all participants, create a medical record file, and record their basic information (gender, age) as well as contact information and medical history information. All participants will undergo a 68Ga-FAPI PET/CT when recurrence or metastasis is suspected. The imaging response measurements will be compared with follow-up results or histopathological findings as the gold standard.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with thyroid cancer who have undergone surgery and are suspected of recurrence or metastasis during clinical evaluation.
2. Signed and dated informed consent form.
3. Commitment to comply with research procedures and co-operation in the implementation of the full research process.
4. Aged 18-80 years old.

Exclusion Criteria:

1. Patients with serious illnesses that researchers consider unsuitable for participation in this clinical study. Such as severe heart and lung failure, severe bone marrow suppression, severe liver and kidney dysfunction, etc.
2. Intestinal perforation, complete intestinal obstruction.
3. Pregnant women and women who may be pregnant, women who are breastfeeding.
4. Non-compliant person.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients and outpatients at Ruijin Hospital who meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of recurrent or metastatic thyroid cancer | Within 1 week after enrollment
  The value of 68Ga-FAPI PET/CT in detecting recurrent and metastatic lesions in patients with thyroid cancer after surgery

SECONDARY OUTCOMES:
Standardized uptake value(SUV) | Within 1 week after enrollment
  SUV of 68Ga-FAPI uptake on PET/CT images for tumor lesions
Disease free survival | 3 years
  Disease free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital affiliated to Shanghai Jiao Tong University of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No